CLINICAL TRIAL: NCT03613480
Title: Study of Quality of Life in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Quality of Life in Non-alcoholic Fatty Liver Disease (QOLNAFLD)
Acronym: QOLNAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Christos Triantos, Assistant Professor in Internal Medicine and Gastroenterology, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 328/15.05.2018
Record Dates: First submitted 2018-05-17; First posted 2018-08-03 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: All eligible patients will be randomized to receive either counseling sessions or care as usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Patients will receive 6 brief (20-30mins) counseling sessions based on the principles of Motivational Interviewing by a trained member (psychiatrist) of the research team. The first session will take place at 2 weeks after baseline and the following 5 sessions will be conducted at a monthly basis.
  Interventions: Other: Motivational Interviewing
- Care as usual (No Intervention): Patients will be followed-up by the hepatologists of the Outpatient Department at regular time intervals and will be re-evaluated after 6 months from baseline

INTERVENTIONS:
Other: Motivational Interviewing — Regular sessions of Motivational Interviewing at 2 weeks and then at monthly intervals for a period of 6 months
  Arms: Motivational Interviewing

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a highly prevalent disorder which is directly linked to lifestyle patterns and is associated with poor quality of life, increased fatigue and psychological distress. The aim of the current study is to evaluate quality of life, fatigue and psychological functioning in NAFLD patients and assess the impact of systematic counseling on patients' psychosocial functioning.

DETAILED DESCRIPTION:
Introduction: The term non-alcoholic fatty liver disease (NAFLD) encompasses a spectrum of disorders ranging from simple steatosis to steatohepatitis, in the absence of other known causes of liver steatosis. NAFLD is a highly prevalent disorder which is directly linked to patients' lifestyle and is accompanied by severe co-morbidities. Although there is a wealth of studies on NAFLD's pathogenesis, natural course and treatment, few investigations have focused on patients' quality of life (QoL) and even fewer have evaluated the impact of therapeutic interventions on patients' quality of life and psychosocial functioning. In this context, there is a significant literature gap, given that modern research and clinical practice should aim at meeting patients' subjective physical and psychosocial needs and improving their overall quality of living.

Aim-Methods: In this context, the aim of the present study is to assess the effect of systematic counseling on NAFLD patients' quality of life, psychological distress, fatigue and lifestyle habits.

The current study will be conducted at the Gastroenterology Department of the University Hospital of Patras with the collaboration of the Department of Psychiatry. NAFLD patients will be invited to enrol to the study after being thoroughly informed about its aim and methods. Eligible patients will be assessed at baseline and then will be randomized to receive either systematic counseling based on the principles of Motivational Interviewing or care as usual. All participants will be re-evaluated at 6 months after study initiation. In addition, all patients will be submitted to laboratory tests including complete blood count, serum albumin, hemoglobin, gamma-globulin, ALT, AST, γGT, ALP, bilirubin, PT, INR, urea, creatinine, total cholesterol, LDL, HDL, triglycerides both at baseline and at study completion

ELIGIBILITY:
Inclusion Criteria:

• Non-alcoholic fatty liver disease according to the EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease

Exclusion Criteria:

* Chronic viral hepatitis or any other severe chronic liver disease
* Major psychopathology
* Severe cognitive or neurological deficits
* Cancer or any other severe chronic disease not associated with NAFLD
* Inadequate knowledge of the Greek language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Health Survey 36 Short Form (SF36) | 6 months
  The SF36 is a self-report, generic quality of life instrument, which includes eight multi-item scales (36 items) that evaluate the extent to which an individual's health limits his or her physical, emotional, and social well-being. The SF-36 covers eight domains of HRQOL, namely physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems, and mental health. Scores on each subscale range from 0 to 100, with higher scores indicating a better quality of life. Sub-scales scores are calculated according to an algorithm described in the SF36 manual.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  This is a psychometric tool measuring psychological distress. It is comprised of 14 items, 7 items for anxiety and 7 items for depression. Each item is scored from 0 to 3 and subscale scores are calculated by summing the 7 item scores. Each subscale ranges from 0-21 and higher scores indicate greater severity of depressive and anxious symptoms
Chronic Liver Disease Questionnaire (CLDQ) | 6 months
  This is a disease-specific instrument measuring quality of life. It encompasses 29 items contained within six domains including abdominal symptoms, fatigue, systemic symptoms, activity, emotional function and worry. A Likert scale response format is used for all items ranging from 1 (most impairment) to 7 (least impairment). Scoring of the questionnaire is performed by dividing each domain score by the number of items per domain.Overall CLDQ score is obtained by adding scores for each item and dividing by the total number of items.
Fatigue Severity Scale | 6 months
  This 9-item scale measures the severity of fatigue and its effect on a person's activity and lifestyle in patients with various disorders. Each item is scored on a 7 point scale with 1=strongly disagree and 7=strongly agree. Total score is calculated by adding each item score. Scores range from 9 to 63 and higher scores indicate greater fatigue severity

SECONDARY OUTCOMES:
Alanine aminotransferase levels (ALT) | 6 months
  This is a blood test measuring the serum concentration of alanine aminotransferase which is elevated in liver damage. ALT reference rates range between 20 to 60 IU/L
Aspartate aminotransferase levels (AST) | 6 months
  This is a blood test measuring the serum concentration of aspartate aminotransferase which is elevated in liver damage. AST reference rates range between 5 to 40 IU/L
Body Mass Index (BMI) | 6 months
  The Body Mass Index is a measure of obesity. It is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.Normal BMI ranges from 18.5-24.9

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: No